CLINICAL TRIAL: NCT05198687
Title: Comparison Between Three Different Treatment Modalities for Atrophied Distal Extension Maxillary Ridges Clinical and Radiographic Study
Brief Title: Different Treatment Modalities for Atrophied Distal Extension Maxillary Ridges
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M06030320
Record Dates: First submitted 2021-09-24; First posted 2022-01-20 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2021-09

CONDITIONS: Partial Edentulism Class 1

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- overdentures (Active Comparator): implant overdentures
  Interventions: Procedure: Long implant and partial overdentures; Device: Partial overdentures
- sinus lift (Active Comparator): sinus lift and long implants and screw-retained prosthesis
  Interventions: Procedure: Sinus lift and long implant; Device: Metal ceramic prosthesis on long implants
- short implants (Active Comparator): short implants and screw-retained prosthesis
  Interventions: Procedure: short implant without sinus lift; Device: Metal ceramic prosthesis on short implants

INTERVENTIONS:
Procedure: Long implant and partial overdentures — insertion of long implants anterior to the maxillary sinus to retain partial overdentures
  Arms: overdentures
Procedure: Sinus lift and long implant — performing sinus lift surgical procedure with simultaneous placement of long implants to support screw-retained prosthesis
  Arms: sinus lift
Procedure: short implant without sinus lift — placement of short implants in the remaining bone above maxillary sinus to support screw-retained prosthesis without performing sinus lift
  Arms: short implants
Device: Partial overdentures — Distal extension metallic partial dentures retained by attachments to the implants
  Arms: overdentures
Device: Metal ceramic prosthesis on long implants — porcelain fused to metal fixed screw-retained prosthesis supported by long implants
  Arms: sinus lift
Device: Metal ceramic prosthesis on short implants — porcelain fused to metal fixed screw-retained prosthesis supported by short implants
  Arms: short implants

SUMMARY:
This study will compare clinical and radiographic outcomes of three different treatment modalities for atrophied distal extension maxillary ridges these modalities include

1. Implant retained distal extension RPD
2. Sinus lift and long implant and screw-retained prosthesis
3. Short implant and screw-retained prosthesis

DETAILED DESCRIPTION:
Patient selection:

For this study, 60 patients were selected from the clinic of Prosthodontic Department, Faculty of Dentistry, Mansoura University.

Inclusion criteria:

The patients will be selected according to the following:

* They have distal extension maxillary ridge with sinus pneumatization and remaining alveolar bone height 6- 8mm as verified by preoperative CBCT, have no previous denture experience. They are healthy, free from any systemic diseases relating to the bone resorption (diabetes - hyperparathyroidism). This can be achieved through medical history and clinical examination by a physician and laboratory investigations.
* Posterior maxillary alveolar ridge deficient in height, width and covered with healthy firm mucosa.
* Patients are less satisfied with conventional RPD.
* Absence of maxillary sinus diseases. Exclusion criteria

Patients were not eligible for this work if any of the following criteria were met:

* Acute or chronic sinus pathology
* History of a sinus augmentation in the past in the relevant sinus
* Poor dental hygiene. Smoker.
* Compromised general health (uncontrolled diabetes, bleeding disorder….). All patient were informed about all procedures that will be done and they sign the written consent form of ethical committee in faculty of dentistry Mansoura university.

Three treatment groups will be classified randomly, as follow:

* Group A: patients received two implant in premolar area mesial to maxillary sinus and used to retain partial overdenture
* Group B: patient underwent sinus lift and receive screw retained prosthesis on long implant
* Group C: patients received short implants in premolar area mesial to maxillary sinus and received screw retained prothesis All implants were inserted using computer guided implant surgery and conventional loading protocol was used.

Evaluation methods Clinical and radiographic evaluation

1. Modified Plaque index. Assessment of plaque accumulation with a modified plaque index (mPI): Score 0: No detection of plaque, Score 1: Plaque only recognized by running a probe across the smooth marginal surface of the implant, Score 2 Plaque can be seen by a naked eye, Score 3 Abundance of soft matter.
2. Gingival index. Assessment of bleeding tendency with a modified sulcus bleeding index (mBI): Score 0 No bleeding when a periodontal probe is passed along the gingival margin adjacent to the implant. Score 1 Isolated bleeding spot visible, Score 2 Blood forms a confluent red line on margin, Score 3 Heavy or profuse bleeding.
3. Attachment level. Distance from the junction implant/crown to the most apically probeable portion, in millimeters.
4. Pocket depth. Distance between the gingival margin and the most apically probable portion, in millimeters Assessed by insertion of a standard periodontal probe with a point diameter of 0.5 mm using a probing force of 0.5 N.
5. Implant stability quotient. Using resonance frequency analysis

   b- Radiographic evaluation will be performed in terms of:

   Vertical bone loss (VBL) will be evaluated as follows:

   The distance between implant plate form and first bone to implant contact (DIM) will be evaluated at T0, T6 and T12. VBL will be calculated by subtracting DIM at T6 and T12 from DIM at T0.

ELIGIBILITY:
Inclusion Criteria:

The patients will be selected according to the following:

* They have distal extension maxillary ridge with sinus pneumatization and remaining alveolar bone height 6- 8mm as verified by preoperative CBCT, have no previous denture experience. They are healthy, free from any systemic diseases relating to the bone resorption (diabetes - hyperparathyroidism). This can be achieved through medical history and clinical examination by a physician and laboratory investigations.
* Posterior maxillary alveolar ridge deficient in height, width and covered with healthy firm mucosa.
* Patients are less satisfied with conventional RPD.
* Absence of maxillary sinus diseases.

Exclusion Criteria:

* Acute or chronic sinus pathology
* History of a sinus augmentation in the past in the relevant sinus
* Poor dental hygiene. Smoker.
* Compromised general health (uncontrolled diabetes, bleeding disorder

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
Plaque index | one year
  measuring plaque accumulation around implants using scores
Gingival index | one year
  measuring gingival inflammation around implants using scores
Probing depth | one year
  measuring peri-implant probing depth in mm
implant stability | one year
  measuring the mobility of the implants using resonance frequency analysis Implant stability quotient)
Marginal bone loss | one year
  measuring crestal bone loss around implants in mm
Patient satisfaction using VAS questionnaire (visual analogue scale) | one year
  Regarding VAS, participants were asked to score their answer according to the amount of satisfaction on a 100mm line (Score zero = no satisfaction at all and score 100 = complete satisfaction). The questions cover several items related to prosthesis such as: retention, stability, comfort, ease of cleaning, ease of speaking, ease of chewing, limited activities due to embarrassment, quality of bolus and appearance.

SECONDARY OUTCOMES:
Prosthetic Aspects | one year
  measuring the incidence of prosthetic aspects and maintenance requirements
Muscle activity | one year
  measure muscles activity in amplitude using electromyographs
maximum bite force | one year
  measuring maximum bite force in newton using bite force transducers

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Mansoura University, Al Mansurah, Eldakahlia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol